CLINICAL TRIAL: NCT03856957
Title: Serrated Lesions Detection With Endocuff-assisted Colonoscopy - A Randomized Controlled Trial
Brief Title: Serrated Lesions Detection With Endocuff-assisted Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Beatriz Ângelo (Other)
Responsible Party: Principal Investigator, Alexandre Ferreira, Dr, Hospital Beatriz Ângelo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0304
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Serrated Lesion; Adenoma; Colorectal Cancer
Keywords: Serrated Lesion; Endocuff; Detection
MeSH Terms: conditions — Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocuff colonoscopy (Experimental): Colonoscopy performed with Endocuff
  Interventions: Device: Endocuff colonoscopy
- Conventional colonoscopy (Placebo Comparator): Colonoscopy performed without any device
  Interventions: Device: control

INTERVENTIONS:
Device: Endocuff colonoscopy — Colonoscopy performed with Endocuff for mucosal inspection and interventions (eg. polypectomy).
  Arms: Endocuff colonoscopy
Device: control — colonoscopy without endocuff
  Arms: Conventional colonoscopy

SUMMARY:
Colorectal cancer (CRC) is a leading cause of morbidity and mortality worldwide, especially in Western countries. CRC is currently considered a preventable disease and screening has been endorsed by several societies, since it has been shown that screening and surveillance are effective in reducing both CRC incidence and mortality. However, recently, concern has risen regarding colonoscopy effectiveness, especially in the right colon. The most accepted explanation for this effectiveness variability is attributed to sessile serrated lesions (SSL), which are more frequent in the proximal colon, more difficult to detect because of their flat morphology and associated with interval CRC, which is the occurrence of CRC after screening colonoscopy and before the next scheduled procedure. Several techniques are emerging to increase the sensitivity of colonoscopy for pre-cancerous lesions, especially adenomas. Recently an endoscopic cap, the Endocuff, was developed to improve adenoma detection. Several studies demonstrated improved adenoma detection with Endocuff-assisted colonoscopy when compared with conventional colonoscopy. Still, the available data for its' role in detecting SSL is very limited. The aim of this randomized controlled trial is to evaluate the effectiveness of Endocuff-assisted colonoscopy in detection of colorectal SSL.

ELIGIBILITY:
Inclusion Criteria:

- Outpatients undergoing elective colonoscopies

Exclusion Criteria:

* Known polyposis syndromes
* Personal colorectal cancer history
* Previous colorectal surgery
* Severe diverticulosis
* Colonic stricture
* Inflammatory bowel disease
* Primary sclerosing cholangitis
* Pregnancy and breastfeeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Average number of serrated lesions ≥ 10 mm detected per colonoscopy | immediate
  Average number of serrated lesions ≥ 10 mm detected per colonoscopy

SECONDARY OUTCOMES:
Serrated lesions detection rate | immediate
  Number of patients with at least one serrated lesion/total number of participants
Average number of serrated lesions < 10 mm detected per colonoscopy | immediate
  Average number of serrated lesions < 10 mm detected per colonoscopy
Average number of adenomas detected per colonoscopy | immediate
  Average number of adenomas detected per colonoscopy
Adenoma detection rate | immediate
  Number of patients with at least one adenoma/total number of participants
Adenocarcinoma detection rate | immediate
  Number of patients with at least one adenocarcinoma/total number of participants
Cecal intubation rate | immediate
  Proportion of colonoscopies with cecal intubation x100
Cecal incubation time | immediate
  time from the rectum to cecum in minutes
Withdrawal time | immediate
  time from the cecum to the rectum in minutes
Incidence of procedure related adverse events | immediate
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beatriz Ângelo, Lisbon, Loures, Portugal